CLINICAL TRIAL: NCT06530147
Title: Comparison Of The Effectiveness Of Transversalis Fascia Plane Block And Transversus Abdominis Plane Block For Postoperative Analgesia After Pediatric Lower Abdominal Surgeries
Brief Title: Transversalis Fascia Plane Block vs Transversus Abdominis Plane Block In Pediatric Surgeries
Status: Completed | Type: Observational
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Hasibe Irban, Principal Investigator, Kocaeli University
Other Study IDs: KAEK/06.bl.02
Record Dates: First submitted 2024-07-05; First posted 2024-07-31 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Postoperative Analgesia
Keywords: Regional anaesthesia; Transversus Abdominis Plane Block; Transversalis Fascia Plane Block; Pediatric Lower Abdominal Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transversalis Fascia Plane Block: One-side ultrasound (US)-guided Transversalis fascia plane (TFP) block with 0.25% bupivacaine will performe after placement laryngeal mask airway before surgery.
  Interventions: Other: Transversalis Fascia Plane Block
- Transversus Abdominis Plane Block: One-side ultrasound (US)-guided Transversus abdominis plane (TAP) block with 0.25% bupivacaine will performe after placement laryngeal mask airway before surgery.
  Interventions: Other: Transversus Abdominis Plane Block

INTERVENTIONS:
Other: Transversalis Fascia Plane Block — One-side ultrasound (US)-guided Transversalis fascia plane (TFP) block with 0.25% bupivacaine will performe after placement laryngeal mask airway before surgery.
  Groups: Transversalis Fascia Plane Block
Other: Transversus Abdominis Plane Block — One-side ultrasound (US)-guided Transversus abdominis plane (TAP) block with 0.25% bupivacaine will performe after placement laryngeal mask airway before surgery.
  Groups: Transversus Abdominis Plane Block

SUMMARY:
In this study, the investigators compared ultrasound-guided transversalis fascia plane (TFP) block and transversus abdominis plane (TAP) block on postoperative analgesic effect in pediatric abdominal surgeries

DETAILED DESCRIPTION:
After being informed about the study and potential risks, written consent was obtained from all patients. In order to effectively manage postoperative analgesia in patients planned for lower abdominal surgery (inguinal hernia and undescended testicles), patients will begin to be observed after routine anesthesia and block techniques applied to the patients. After these procedures, the block is applied to the patient using the appropriate method, under aseptic conditions and under ultrasound guidance. Intraoperative hemodynamic changes of the patients, intraoperative opioid consumption and bispectral index monitoring values of the patients will be kept throughout the peroperative period. Postoperative follow-ups will be made at 0nd, 1st, 2nd, 4th, 6th, 12th, and 24th hours to evaluate the initial analgesic consumption, need for analgesics types, pain levels, and parental satisfaction. In this way, it is aimed to compare the Transversalis Fascia Plan Block and Transversus Abdominis Plan Block as an effective analgesic application in lower abdominal surgery in children and to show the analgesic method that can be used effectively in postoperative pain management.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist Classification (ASA) I-II patients
* 1-7 aged patients
* patients who scheuled elective lower abdominal surgery (inguinal hernia and undescended testis)

Exclusion Criteria:

* Use of anticoagulants
* Allergy of medications to be used
* Presence of infection the area where the block will be applied
* American Society of Anesthesiologist Classification (ASA) III-IV patients
* The study will not include any vulnerable population, such as those in restraints, those in intensive care and those who are unconscious, and those who cannot give personal consent or impressionable subjects.
* Patients who do not agree to participate in the research, parents/legal guardians
* Patients who were operated on with a different incision than planned for any reason.

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients aged between 1 and 7 years who will undergo abdominal surgery will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2024-08-06 (Actual)

PRIMARY OUTCOMES:
Pain scores | at the 6th postoperative hou
  Our primary aim to compare the effect of both blocks groups on the FLACC (Face, Legs, Activity, Cry, Consolability) pain scores at the 6th postoperative hour. FLACC pain scale, zero is designated as the lowest pain level, and ten as the highest pain level.

SECONDARY OUTCOMES:
Pain scores | During postoperative 24 hours
  Secondary objectives will include comparison of patient FLACC (Face, Legs, Activity, Cry, Consolability) pain scores in 24-hour observations of patients. FLACC pain scale, zero is designated as the lowest pain level, and ten as the highest pain level.
Need for analgesic | During postoperative 24 hours
  It should be recorded whether there is a need for analgesics.
Nause and vomiting | During postoperative 24 hours
  The presence or absence of nausea and vomiting symptoms will be recorded.
Parents satisfaction | During postoperative 24 hours
  Parental satisfaction was assessed on a scale ranging from 1 to 5 points parents satisfaction with the applied analgesia methods was evaluated on a scale from 1, indicating the lowest satisfaction, to 5, indicating the highest satisfaction.
Time elapsed until the first analgesic requirement | During postoperative 24 hours
  What type of analgesic is needed. The time elapsed until the first analgesic requirement was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Can Aksu, Study Director — Kocaeli University
Locations (1):
- Hasibe Irban, Kocaeli, Turkey (Türkiye)

REFERENCES:
- [Derived] Irban H, Aksu C. Comparison of the effectiveness of transversalis fascia plane block and transversus abdominis plane block for postoperative analgesia in pediatric lower abdominal surgeries: prospective, single blinded study. BMC Anesthesiol. 2025 Apr 5;25(1):154. doi: 10.1186/s12871-025-03023-z. PMID 40188032